CLINICAL TRIAL: NCT04009811
Title: A New Membrane Obturator Prothesis Concept for Soft Palate Defects
Acronym: VELOMEMBRANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2018/34
Record Dates: First submitted 2019-06-24; First posted 2019-07-05 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Mouth Neoplasms; Velopharyngeal Insufficiency; Speech Disorders; Deglutition Disorders
Keywords: Randomized controlled trial; Palatal obturators
MeSH Terms: conditions — Mouth Neoplasms; Velopharyngeal Insufficiency; Speech Disorders; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suersen obturator then membraneous obturator (Experimental)
  Interventions: Device: Suersen and membraneous obturators evaluation
- Membraneous obturator then Suersen obturator (Experimental)
  Interventions: Device: Suersen and membraneous obturators evaluation

INTERVENTIONS:
Device: Suersen and membraneous obturators evaluation — The patient will wear one month each obturator prothesis (Suersen and membraneous obturators). The order of evaluation will be randomized in two arms.
  Half of patient will first wear one month the membranous obturator then one month the Suersen, the other half of patient will first wear one month the Suersen obturator and one month the membranous obturator.

SUMMARY:
When soft palate defects lead to palatal insufficiency, the patient's quality of life is affected by difficulties swallowing, hypernasality, and poor intelligibility of speech. If immediate surgical reconstruction is not an option, the patient may benefit from the placement of a rigid obturator prosthesis. Unfortunately, the residual muscle stumps are often unable to adequately move this stiff and inert obturator to properly restore the velopharyngeal valve function. The objective of this case report was to describe the use of a membrane obturator prosthesis that incorporates a dental dam to compensate for the soft palate defect.

DETAILED DESCRIPTION:
The velopharyngeal sphincter seals the oropharynx from the nasopharynx during swallowing and speech. This three-dimensional muscular valve closes through the synergistic behavior of the soft palate and the lateral and posterior walls of the pharynx. A soft palate defect surgically acquired in the context of oral cancer may impede complete closure and lead to a palatopharyngeal insufficiency. The resultant airflow escape results in hypernasality, poor speech intelligibility, and swallowing problems (such as leakage of foods and fluids into the nasal airways). The best way to rehabilitate and restore chewing and swallowing is one of the top ten research priorities in head and neck cancer. When the velopharyngeal function cannot be immediately restored with surgical reconstruction, patients can benefit from an obturator prosthesis. This obturator is a rigid extension of acrylic resin positioned at the level of the hard palate that provides surface contact for the remaining musculature. Often, the residual muscle stumps cannot move adequately around this stiff and inert obturator to properly restore the velopharyngeal valve function. The resulting blockage, or free space between the tissues and obturator, is a main cause of prosthetic failure. Subsequently, in many cases, oral functions remain impaired, with a negative impact on the patient's quality of life.

The compensating treatment consists of a provisional removable partial denture (RPD) with a membrane obturator. The membrane consisted of a thick dental dam shaped with scissors to create a 10-mm overlap with the pharyngeal walls that was then perforated with four holes using punch pliers.

The follow-up ends after the last visit. However, our team can provide cares of any patient seeking for dental care, prosthetic treatments and routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 year-old
* Acquired loss of velar or palato-velar substance (maxillectomies of Class I and II a-d, Brown 2010) following the excision of a tumor
* Indication of Suersen obturator prosthesis rehabilitation
* Possible dental rehabilitation with removable prosthesis (retention and stability prosthetic provided without the use of glue, mouth opening allowing fingerprints, presence of saliva, dexterity allowing the insertion and removal of prostheses, as well as the cleaning of devices)
* Having given their consent to participate in the study
* Speaking French, knowing how to read it
* Available and motivated for regular follow-up during the study period

Exclusion Criteria:

* Child under 18
* Allergy to acrylic resin
* Radiotherapy or chemotherapy in progress
* Surgery of the veil programmed during the 3 months necessary for the realization and the wearing of the prostheses.
* Loss of congenital or traumatic palato-velar substance
* Maxillectomies including orbital floor or total maxillectomy
* Pregnant or lactating woman
* Participation in another interventional study
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index (VHI) overall score | Visit M2 : one month after first obturator supply i.e. two months after inclusion
  Min : 0 = Non handicap to Max : 120 = voice handicap maximum
Voice Handicap Index (VHI) overall score | Visit M3 : one month after second obturator supply i.e. three months after inclusion
  Min : 0 = Non handicap to Max : 120 = voice handicap maximum

SECONDARY OUTCOMES:
Deglutition Handicap Index (DHI) overall score | Visit M1 : one month after inclusion
  Min : 0 = Non handicap to Max : 120 = deglutition handicap maximum
Deglutition Handicap Index (DHI) overall score | Visit M2 : two months after inclusion
  Min : 0 = Non handicap to Max : 120 = deglutition handicap maximum
Deglutition Handicap Index (DHI) overall score | Visit M3 : three months after inclusion
  Min : 0 = Non handicap to Max : 120 = deglutition handicap maximum
Health-related quality of life EORTC QLQ-C30 questionnaire score | Visit M1 : one month after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life
Health-related quality of life EORTC QLQ-C30 questionnaire score | Visit M2 : two months after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life
Health-related quality of life EORTC QLQ-C30 questionnaire score | Visit M3 : three months after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life
Head and Neck quality of life EORTC QLQ-H&N35 questionnaire score | Visit M1 : one month after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life
Head and Neck quality of life EORTC QLQ-H&N35 questionnaire score | Visit M2 : two months after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life
Head and Neck quality of life EORTC QLQ-H&N35 questionnaire score | Visit M3 : three months after inclusion
  Min : 0 = lower level of quality of life to Max : 100 = better level of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARRIVE, DDS, Study Chair — Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique (USMR) du CHU de Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naveau A, Kret M, Plaire V, Delorme O, Marchi S, de Bataille C, Destruhaut F, Arrive E, Bou C. Efficacy of a new membrane obturator prosthesis in terms of speech, swallowing, and the quality of life of patients with acquired soft palate defects: study protocol of the VELOMEMBRANE randomized crossover trial. Trials. 2022 Mar 18;23(1):221. doi: 10.1186/s13063-022-06163-6. PMID 35303932